CLINICAL TRIAL: NCT03705104
Title: Living Well with Chronic Pain: Using Person-centered E-health Design to Support Self-management
Brief Title: Living Well with Chronic Pain
Acronym: EPIO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: The Research Council of Norway (Other); University of Oslo (Other); University College of Southeast Norway (Other); Diakonhjemmet Hospital (Other); Vestre Viken Hospital Trust (Other); Drammen municipality, Norway (Unknown); Mayo Clinic (Other); University of Twente (Other); University of Washington (Other); University of Florida (Other)
Responsible Party: Principal Investigator, Lise Solberg Nes, Center Director, Head of Research, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018/799
Record Dates: First submitted 2018-09-20; First posted 2018-10-15 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Chronic Pain, Widespread
Keywords: Pain; Chronic Pain; Self-management; E-health; Appication; App; Intervention; Cognitive Behavioral Therapy; CBT; Acceptance and Commitment Therapy; ACT; Psychological well-being
MeSH Terms: conditions — Chronic Pain; Pain; Alzheimer Disease; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- EPIO (e-health intervention) (Experimental): Participants will get access to one module every third day (total 9 modules). The app consists of cognitive behavioral pain self-management material, including educational material and relaxation training exercises.
  Interventions: Behavioral: EPIO
- treatment as usual (No Intervention): Participants will get treatment as usual during the study. All participants will get access to the app after ended study if interested.
- Experimental without introduction group and follow up phone calls (Active Comparator): One extra arm (non randomized) has been included to examine whether participants who receive the EPIO intervention without receiving an introduction session and follow up phone calls will still describe benefiting from the receiving the intervention
  Interventions: Behavioral: EPIO

INTERVENTIONS:
Behavioral: EPIO — App for self-management of chronic pain An app consisting of 9 modules focusing on cognitive behavioral pain self-management.
  Other Names: e-health intervention for chronic pain
  Arms: EPIO (e-health intervention); Experimental without introduction group and follow up phone calls

SUMMARY:
The goal of this project is to test the effect of an interactive e-health intervention for people with chronic pain.

DETAILED DESCRIPTION:
Chronic pain conditions are common and difficult to cure. As much as 30% of adults in Norway experience moderate-to-severe chronic pain, i.e., pain having lasted more than 3 months. Chronic pain is also the most common cause of sick leave and disability pension in Norway. Despite a clear request from the authorities, e-health interventions for chronic pain has not yet been tested and implemented.

The aim of this study is to investigate the effect of an interactive e-health intervention for people living with chronic pain, using outcome measures such as pain intensity, pain acceptance, anxiety/depression and quality of life.

The e-health intervention will first be tested in a pilot study with 50 patients with different pain diagnoses and eventually in a randomized controlled trial with a sample of 240 patients with different pain diagnoses. The intervention will consist of one face-to-face introductory group followed by 9 app-based modules containing cognitive behavioral pain self-management material. The 9 modules will be distributed over minimum 27 days (minimum 3 days per module). The participants in the randomized controlled trial will be randomly assigned to use the e-health intervention or to a treatment as usual control group. Both groups will receive outcome measures to complete at baseline and at 3, 6 and 12 months.

Post-RCT, the EPIO study will also include a non-randomized group receiving the app-based EPIO program but without receiving an introduction session and follow up phone calls to examine potential benefits from receiving the app-based program only.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain (pain > 3 months)
* > 18 years of age
* Able to write/read/speak Norwegian
* Have their own smart phone, PC or tablet

Exclusion Criteria:

* Cancer related pain
* Migraine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2019-12-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory (BPI) (Short Form) - Assessing change | Baseline, and at 3, 6, and 12 months.
  9 item scale measuring pain interference on function. Using this measure, respondents rate their worst, least, average, and current pain intensity and also rate the degree to which pain interferes with 7 domains of functioning (general activity, mood, walking ability, normal work, relations with other persons, sleep, and enjoyment of life) on a scale of 0 to 10.
  There is no scoring algorithm, but "worst pain" or the arithmetic mean of the four severity items can be used as measures of pain severity; the arithmetic mean of the seven interference items can be used as a measure of pain interference.

SECONDARY OUTCOMES:
Pain Catastrophizing Scale (PCS) - Assessing change | Baseline, and at 3, 6, and 12 months.
  13 item scale measuring helplessness, magnification and rumination. Patients rate items on a scale from 0 (not at all) to 4 (all the time). The total score range for the PCS is 0 to 52, with higher scores reflecting higher degrees of catastrophizing.
Chronic Pain Acceptance Questionnaire (CPAQ) - Assessing change | Baseline, and at 3, 6, and 12 months.
  8 item scale measuring pain acceptance. It is scored on a 7-point Likert scale (0 = never true; 6 = always true). Higher scores reflect higher acceptance of pain.
Self-Regulatory Fatigue 18 (SRF-18) - Assessing change | Baseline, and at 3, 6, and 12 months.
  18 item scale measuring self-regulatory capacity with cognitive, emotional, and behavioral components. Items are scored on a 5-point Likert scale (1 to 5). The obtainable score range is 18 to 90, with higher numbers reﬂecting higher SRF.
The Hospital Anxiety and Depression Scale (HADS) - Assessing change | Baseline, and at 3, 6, and 12 months.
  14 item scale measuring anxiety and depression. Respondents are asked to indicate which of 4 response options (rated from 0-3; score range, 0-42) comes closest to describing how they have been feeling in the previous week for each item. Scores from 0-7 on the subscales are regarded as being in the normal range; a score of 11 or higher indicates a probable presence of a mood disorder, and a score of 8-10 is suggestive of the presence of the state.
System Usability Scale (SUS) | At 3 months
  1o item scale measuring usability, with five response options for respondents; from Strongly agree to Strongly disagree. The obtainable score range is 25 to 100. A SUS score above a 68 would be considered above average and anything below 68 is below average.
RAND Health Related Quality of Life - Assessing change | Baseline, and at 3, 6, and 12 months.
  36 item scale measuring health related quality of life. The RAND-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.

CONTACTS AND LOCATIONS:
Overall Officials: Lise Solberg Nes, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bostrom K, Borosund E, Eide H, Varsi C, Kristjansdottir OB, Schreurs KMG, Waxenberg LB, Weiss KE, Morrison EJ, Stavenes Stole H, Cvancarova Smastuen M, Stubhaug A, Solberg Nes L. Short-Term Findings From Testing EPIO, a Digital Self-Management Program for People Living With Chronic Pain: Randomized Controlled Trial. J Med Internet Res. 2023 Aug 25;25:e47284. doi: 10.2196/47284. PMID 37624622
- [Derived] Bostrom K, Varsi C, Eide H, Borosund E, Kristjansdottir OB, Schreurs KMG, Waxenberg LB, Weiss KE, Morrison EJ, Nordang EF, Stubhaug A, Nes LS. Engaging with EPIO, a digital pain self-management program: a qualitative study. BMC Health Serv Res. 2022 Apr 29;22(1):577. doi: 10.1186/s12913-022-07963-x. PMID 35488295
- [Derived] Eiken AG, Nordanger DO, Solberg Nes L, Varsi C. Patients' Experiences of Using an eHealth Pain Management Intervention Combined With Psychomotor Physiotherapy: Qualitative Study. JMIR Form Res. 2022 Mar 16;6(3):e34458. doi: 10.2196/34458. PMID 35293866
- [Derived] Varsi C, Ledel Solem IK, Eide H, Borosund E, Kristjansdottir OB, Heldal K, Waxenberg LB, Weiss KE, Schreurs KMG, Morrison EJ, Stubhaug A, Solberg Nes L. Health care providers' experiences of pain management and attitudes towards digitally supported self-management interventions for chronic pain: a qualitative study. BMC Health Serv Res. 2021 Mar 25;21(1):275. doi: 10.1186/s12913-021-06278-7. PMID 33766028
- [Derived] Bostrom K, Borosund E, Varsi C, Eide H, Flakk Nordang E, Schreurs KM, Waxenberg LB, Weiss KE, Morrison EJ, Cvancarova Smastuen M, Stubhaug A, Solberg Nes L. Digital Self-Management in Support of Patients Living With Chronic Pain: Feasibility Pilot Study. JMIR Form Res. 2020 Oct 23;4(10):e23893. doi: 10.2196/23893. PMID 33094734
- [Derived] Ledel Solem IK, Varsi C, Eide H, Kristjansdottir OB, Borosund E, Schreurs KMG, Waxenberg LB, Weiss KE, Morrison EJ, Haaland-Overby M, Bevan K, Zangi HA, Stubhaug A, Solberg Nes L. A User-Centered Approach to an Evidence-Based Electronic Health Pain Management Intervention for People With Chronic Pain: Design and Development of EPIO. J Med Internet Res. 2020 Jan 21;22(1):e15889. doi: 10.2196/15889. PMID 31961331
- [Derived] Ledel Solem IK, Varsi C, Eide H, Kristjansdottir OB, Mirkovic J, Borosund E, Haaland-Overby M, Heldal K, Schreurs KM, Waxenberg LB, Weiss KE, Morrison EJ, Solberg Nes L. Patients' Needs and Requirements for eHealth Pain Management Interventions: Qualitative Study. J Med Internet Res. 2019 Apr 1;21(4):e13205. doi: 10.2196/13205. PMID 30877780
- See also: Study web page — http://epio.no